CLINICAL TRIAL: NCT06651840
Title: Comparison Between Coblation Versus Bipolar Diathermy in Management of Refractory Idiopathic Recurrent Anterior Epistaxis in Children.
Brief Title: Coblation Versus Bipolar Diathermy in Management of Refractory Idiopathic Recurrent Anterior Epistaxis in Children.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Hosni Anwar Mejalli, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Coblation in child's epistaxis
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Epistaxis Nosebleed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: patients in this group will be managed with bipolar diathermy "Standard technique". (Active Comparator): The bipolar technique for group A:
  A bipolar with straight blade will be used with a footplate-operated switch to control the coagulation time, and the length, width and depth of penetration of the thermal power.
  The lesion will be coagulated in a distal-to-proximal direction to achieve a uniform gray-white coagulation zone in the lesion and surrounding tissue. Multiple ablations at the same area should be avoided to avoid septal perforation. After finishing coagulation small gauze impregnated with antibiotic ointment will be applied for 2 hours postoperatively.
  Interventions: Procedure: bipolar diathermy "Standard technique".
- Group B: patients in this group will be managed with coblation technique. (Experimental): The coblation technique for group B:
  An coblator with tonsillar blade will be used with a footplate-operated switch to control the coagulation time, and the length, width and depth of penetration of the thermal power.
  The lesion will be coagulated in a distal-to-proximal direction to achieve a uniform gray-white coagulation zone in the lesion and surrounding tissue. Multiple ablations at the same area should be avoided to avoid septal perforation. After finishing coagulation small gauze impregnated with antibiotic ointment will be applied for 2 hours postoperatively.
  Interventions: Procedure: coblation technique.

INTERVENTIONS:
Procedure: bipolar diathermy "Standard technique". — The bipolar technique for group A:
  A bipolar with straight blade will be used with a footplate-operated switch to control the coagulation time, and the length, width and depth of penetration of the thermal power.
  The lesion will be coagulated in a distal-to-proximal direction to achieve a uniform gray-white coagulation zone in the lesion and surrounding tissue. Multiple ablations at the same area should be avoided to avoid septal perforation. After finishing coagulation small gauze impregnated with antibiotic ointment will be applied for 2 hours postoperatively.
  Arms: Group A: patients in this group will be managed with bipolar diathermy "Standard technique".
Procedure: coblation technique. — The coblation technique for group B:
  An coblator with tonsillar blade will be used with a footplate-operated switch to control the coagulation time, and the length, width and depth of penetration of the thermal power.
  The lesion will be coagulated in a distal-to-proximal direction to achieve a uniform gray-white coagulation zone in the lesion and surrounding tissue. Multiple ablations at the same area should be avoided to avoid septal perforation. After finishing coagulation small gauze impregnated with antibiotic ointment will be applied for 2 hours postoperatively.
  Arms: Group B: patients in this group will be managed with coblation technique.

SUMMARY:
The aim of this study is to compare the outcomes of coblation technique versus bipolar technique in management of RAE in children regarding the following:

1. Efficacy of each method to stop bleeding.
2. Technical feasibility.
3. Mucosal healing and crust formation.
4. Post operative complications like: synechia formation and septal perforation.
5. Nostril stenosis/ atresia.

DETAILED DESCRIPTION:
Epistaxis commonly referred to as "nosebleed" remains to be one of the most common ENT emergencies presenting to the accident and emergency departments (AED) worldwide. Idiopathic epistaxis is a common complaint seen in children in rhinology outpatient clinics. In most pediatric cases, idiopathic epistaxis originates from Kiesselbach's plexus, which is located in the anteroinferior portion of the nasal septum; thus, this condition is also known as recurrent anterior epistaxis (RAE). The ideal treatment for idiopathic RAE has yet to be elucidated. In most cases only leaning forwards, pinching of the nose and washing of the face and nose with cold water is all that is needed to stop the epistaxis; in other cases, more aggressive interventions as using nasal packing or chemical cauterization are needed. Although silver nitrate cautery is the most common method of chemical cautery for the treatment of RAE, it has mainly been used to control bleeding associated with small vessels and ulceration of the nasal mucosa . Electrosurgery appears to be more effective than silver nitrate in controlling bleeding telangiectasias. Johnson et al. suggested that bipolar electrocautery may be a superior treatment in children with RAE at risk of severe bleeding, in whom chemical cautery will likely fail. Coblation is a minimally invasive therapeutic technique that can cover a large tissue volume, thus allowing for rapid ablation and a large area of coagulation with minimal side effects. Review of the available literatures doesn't compare between these two methods "Bipolar versus coblation regarding their efficacy to control RAE in children". In this research we will study the outcomes of both techniques.

ELIGIBILITY:
Inclusion Criteria:

1. A history of repeated unilateral epistaxis with at least four episodes, at least one episode per week during the preceding 4 weeks.
2. Age > 5 years of age and < 18 years of age.
3. Failure of topical treatment with an antiseptic ointment, with or without silver nitrate cautery.
4. A Katsanis epistaxis scoring system (ESS) score of 7-10.
5. Bleeding originating from Kiesselbach's plexus, located in the anteroinferior portion of the nasal septum.

Exclusion Criteria:

1. Patients < 5 years of age and >= 18 years of age.
2. Patients with bilateral epistaxis.
3. Patients with bleeding tendencies like: Hemophilia, Leukemia, Idiopathic thrombocytopenic purpura, Von Willebrand disease and Thrombasthenia.
4. Patients with previous nasal surgeries.
5. Patients with hereditary hemorrhagic telangiectasia.
6. Patients with vascular lesions like: angiofibroma, pyogenic granuloma and bleeding polypus.
7. Patients who are unfit for surgery.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successful hemostasis on the day of the procedure. | The first 24 hours postoperative
  No epistaxis within the first 24 hours of the procedure.

SECONDARY OUTCOMES:
Postoperative complications | 6 months
  1. Rate of rebleeding rates at 1 and 4 weeks, and 6 months.
  2. Rate of mucosal healing.
  3. Rate of postoperative crust formation.
  4. Rate of postoperative synechiae formation.
  5. Rate of postoperative septal perforation.

CONTACTS AND LOCATIONS:
Overall Officials: Aly R Selim, Professor, Study Chair — Professor; Shimaa I Abdallah, Ass.Prof, Study Director — Assistant Professor

REFERENCES:
- [Background] Lou ZC. Hemostasis of idiopathic recurrent epistaxis in children with microwave ablation: a prospective pilot case series. J Otolaryngol Head Neck Surg. 2019 Dec 18;48(1):72. doi: 10.1186/s40463-019-0393-0. PMID 31852515